CLINICAL TRIAL: NCT06294574
Title: Improved Successful Retrieval Rate of HydroMARK Plus Breast Biopsy Site Marker in Comparison to HydroMARK as Well as Improved Surgeon Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mammotome (Unknown)
Responsible Party: Principal Investigator, Ceren Yalniz, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300011943; 000544990 (Other Grant/Funding Number: Mammotome)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hydromark plus clip placement (Experimental): Patients with a previously placed HydroMARK T3 coil clip or a clip made by another manufacturer and will have a HydroMARK Plus clip placed during the scout localization procedure for this study. Breast surgeons will perform retrieval and then complete a satisfaction survey to compare the two clips.
  Interventions: Device: HydroMARK Plus Clip

INTERVENTIONS:
Device: HydroMARK Plus Clip — Each patient will undergo a breast localization procedure, and a HydroMARK plus clip will be placed.

SUMMARY:
The purpose of the study is to test how successful the retrieval rate of the new HydroMARK Plus Breast Biopsy Site Marker in comparison to HydroMARK.

DETAILED DESCRIPTION:
Study objectives

Primary objective

Assess the successful retrieval rates of the HydroMARK Plus clip

Secondary objective

Determine the level of satisfaction of the surgeon with the retrieval of the HydroMARK Plus clip

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy clips scheduled for surgery with SCOUT localization

Exclusion Criteria:

* Patients who didn't have surgery, patients younger than 18 years old
* Patients older than 90 years old
* Inmates
* Non-English speakers

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retrieval rate of the HydroMARK Plus clip. | Date of HydroMARK Plus Clip placement to 1 week plus or minus 5 days
  The primary endpoint of HydroMARK Plus retrieval rate will be estimated with % and two-sided 95% CI using normal approximation. A paired McNemar Test will be used to compare HydroMARK Plus retrieval rate and HydroMARK retrieval rate, and the 95% CI for the difference of retrieve rate will be estimated using the Newcombe's Score method.

SECONDARY OUTCOMES:
Level of satisfaction of the surgeon with the retrieval of the HydroMARK Plus clip. | Date of retrieval surgery to 1 week.
  Surgeon satisfaction will be evaluated using a Likert scale survey.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Yalniz, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No